CLINICAL TRIAL: NCT00746759
Title: Airway Epithelium Gene Expression in the Diagnosis of Lung Cancer: AEGIS IDE
Brief Title: Airway Epithelium Gene Expression: AEGIS IDE
Acronym: AEGIS IDE
Status: Completed | Type: Observational
Sponsor: Allegro Diagnostics, Corp. (Industry)
Collaborators: University of Pennsylvania (Other); Columbia University (Other); Temple University (Other); Indiana University (Other); University of Alabama at Birmingham (Other); University of Missouri-Columbia (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of Wisconsin, Madison (Other); Medical University of South Carolina (Other); National Jewish Health (Other); Overlake Hospital Bellevue WA (Unknown); Pulmonary and Allergy Associates of New Jersey (Unknown); Pulmonary Associates of Arizona (Unknown); William Jennings Bryan Dorn VA Medical Center (U.S. Federal Agency); Virginia Commonwealth University (Other); Jamaica Hospital Medical Center (Other); North Florida/South Georgia Veterans Health System (Other); Steward St. Elizabeth's Medical Center of Boston, Inc. (Other); University of California, Davis (Other); Yale University (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ADx-0001: IDE G090194
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Smoker; Former Smoker; Gene Expression; Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cells, Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard of Care
  Interventions: Device: Biomarker (not used as an intervention)

INTERVENTIONS:
Device: Biomarker (not used as an intervention) — This study is an observational study. There is no intervention.
  Other Names: BronchoGen

SUMMARY:
The purpose of the research study is to develop a new, more sensitive, and less invasive test for diagnosing lung cancer at an earlier stage, when it can more easily be cured. The investigators hypothesize that certain genes are expressed differently in current and former smokers who have lung cancer, and this difference in gene expression may be a biomarker for lung cancer.

DETAILED DESCRIPTION:
Allegro Diagnostics is funding this multi-center study to validate and extend a new diagnostic tool measuring global gene expression in airway epithelial cells obtained at routine bronchoscopy in suspect lung cancer patients. The test, which is highly sensitive and specific for lung cancer, measures the levels of expression of genes in cells brushed from the large bronchi during diagnostic bronchoscopy. Similar brushings of epithelial cells from the nose will be analyzed to determine if gene expression in these cells can be used as a screening tool in subjects who may have now or be at risk for developing lung cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients being evaluated for the diagnosis of possible lung cancer or "rule out lung cancer" and undergoing clinically indicated bronchoscopy
* All patients are required to be at least 21 years of age and be able to understand and sign the informed consent form
* Patient must be a current or former cigarette smoker

Exclusion Criteria:

* A pulmonary physician does not recommend that bronchoscopy be performed
* Inability to understand the written consent form and comply with requirements of the study
* History of prior primary lung cancer
* Immediately prior to bronchoscopy, the patient has been on a mechanical ventilator for >24 consecutive hours.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of enrolled medical centers who are undergoing clinically indicated bronchoscopy for suspect lung cancer and who are current or former cigarette smokers.
Sampling Method: Non-Probability Sample
Enrollment: 1331 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Lung Cancer Diagnosis (positive or negative) | 12 months
  Patients may be followed at 12 months post bronchoscopy to finalize diagnosis if diagnosis had not previously been confirmed. The biomarker score will be compared to the standard diagnosis to evaluate the sensitivity, specificity, and negative predictive values of the biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Whitney, PhD, Study Director — Allegro Diagnostics
Locations (21):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - Pulmonary Associates of Arizona, Phoenix, Arizona
  - University of California- Davis, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Yale Univeristy, New Haven, Connecticut
  - North Florida/South Georgia VA, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - LSU, New Orleans, Louisiana
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Pulmonary and Allergy Associates of New Jersey, Summit, New Jersey
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dorn VA, Columbia, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia
  - Overlake Hospital, Bellevue, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Vachani A, Whitney DH, Parsons EC, Lenburg M, Ferguson JS, Silvestri GA, Spira A. Clinical Utility of a Bronchial Genomic Classifier in Patients With Suspected Lung Cancer. Chest. 2016 Jul;150(1):210-8. doi: 10.1016/j.chest.2016.02.636. Epub 2016 Feb 16. PMID 26896702
- [Derived] Silvestri GA, Vachani A, Whitney D, Elashoff M, Porta Smith K, Ferguson JS, Parsons E, Mitra N, Brody J, Lenburg ME, Spira A; AEGIS Study Team. A Bronchial Genomic Classifier for the Diagnostic Evaluation of Lung Cancer. N Engl J Med. 2015 Jul 16;373(3):243-51. doi: 10.1056/NEJMoa1504601. Epub 2015 May 17. PMID 25981554